CLINICAL TRIAL: NCT06623266
Title: Neck Observation Versus Selective Neck Dissection in Patients with CT1N0M0 Oral Squamous Cell Carcinoma: a Multicenter Randomized Controlled Trial
Brief Title: Neck Observation or Elective Neck Dissection in CT1N0M0 OSCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Lai-ping Zhong, Professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Acromion
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-09

CONDITIONS: Oral Cancer; Lymph Node Metastasis
Keywords: Oral squamous cell carcinoma; Early stage; Neck dissection; Neck observation; Lymph node metastasis rate
MeSH Terms: conditions — Mouth Neoplasms; Lymphatic Metastasis; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 to the experimental or control arm. Experimental arm: radical resection of the primary lesion only, with neck observation, the safety margins of the primary lesion are 1.0-1.5cm far away from the palpable margins of the lesion.
  Control arm: radical resection of the primary lesion with 1.0-1.5cm safety margins, and elective neck dissection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Placebo Comparator): The patients in the experimental arm will receive radical resection of the primary lesion only, with neck observation, the safety margins of the primary lesion are 1.0-1.5cm far away from the palpable margins of the lesion. Ultrasonography, CT scan, and/or MRI examination will be used to detect lesions.
  Interventions: Procedure: Neck management
- Control arm (Active Comparator): The patients in the control arm will receive radical resection of the primary lesion with the safety margins of the primary lesion are 1.0-1.5cm far away from the palpable margins of the lesion, they will also receive simultaneous elective neck dissection. Ultrasonography, CT scan, and/or MRI examination will be used to detect lesions.
  Interventions: Procedure: Neck management

INTERVENTIONS:
Procedure: Neck management — In the experimental arm: the neck management is neck observation, simultaneous elective neck dissection is not performed during the surgical resection of primary lesion. The patients will be followed up every two months for at least two years, focusing on the lymph node metastasis and local recurrence. Ultrasonography, CT scan, and/or MRI will be used to detect lesions.
  In the control arm: the neck management is elective neck dissection. Simultaneous elective neck dissection is performed during the surgical resection of primary lesion. The patients will be followed up every two months for at least two years, focusing on the lymph node metastasis and local recurrence. Ultrasonography, CT scan, and/or MRI will be used to detect lesions.

SUMMARY:
To evaluate the clinical outcomes of 2-year lymph node metastasis rate, disease-free survival, overall survival, and health-related quality of life in the patients with cT1N0M0 oral squamous cell carcinoma, who receive primary lesion resection combined with elective neck dissection or primary lesion resection only.

DETAILED DESCRIPTION:
For the patients with cT1N0M0 oral squamous cell carcinoma (OSCC), surgical resection of primary lesion is the preferred treatment. However, there are still debates on the neck management, some surgeons suggest elective neck dissection (END), and some surgeons suggest neck observation (NOB). The advantage of elective neck dissection is to clear the potential occult neck lymph node metastasis (about 15%), which could not be detected by clinical examination and imaging examination, and the disadvantage of END is to cause neck deformity, large scars, stiff neck and shoulders, difficulty in raising shoulders, and increase medical costs. The disadvantage of NOB is the risk of lymph node metastasis and disease progression. However, recent retrospective studies show that END has no potential benefit in improving survival in cT1N0M0 patients. The aim of the present trial is to compare the clinical outcomes between the cT1N0M0 OSCC patients, who receive primary lesion resection combined with elective neck dissection or primary lesion resection only, on the aspects of 2-year lymph node metastasis rate, disease-free survival, overall survival, and health-related quality of life. A total number of 300 patients will be recruited, including 150 patients in the experimental arm and 150 patients in the control arm. Experimental arm: radical resection of the primary lesion only, with neck observation, the safety margins of the primary lesion are 1.0-1.5cm far away from the palpable margins of the lesion. Control arm: radical resection of the primary lesion with 1.0-1.5cm safety margins, and elective neck dissection. A complete medical history will be obtained and tumor assessment will be performed at baseline. Patients will be followed-up by every three months in the first 2 years, every six months in the next 3-5 years, and once a year thereafter until death or data censoring. Two-year lymph node metastasis rate, disease-free survival, overall survival, and health-related quality of life will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Tumor site: tongue, gingiva, buccal mucosa, floor of mouth, hard palate, retromolar eara
* Clinical stage is cT1N0M0 (AJCC 8th edition)
* Pathological diagnosis of squamous cell carcinoma
* Sign the informed consent form

Exclusion Criteria:

* More than 2 lesions found in the oral cavity
* Known history of malignant tumor within five years (unless the patient has undergone curative treatment and there is no disease recurrence within 5 years since the start of treatment)
* History of unilateral or bilateral neck dissection in the past
* History of previous head and neck radiotherapy
* Pregnant or lactating women
* Severe, uncontrolled infection or known HIV infection; or previous organ transplantation, stem cell or bone marrow transplantation
* Participated in other clinical studies within 30 days before enrollment
* Other circumstances that the researcher considers unsuitable for participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of 2-year lymph node metastasis | 2 years
  Lymph node metastasis is confirmed by pathological examinations, using fine needle aspiration cytology or biopsy. The rate of 2-year lymph node metastasis rate is reported as the percentage of patients who are free from lymph node metastasis for 2 years from the date of randomization.

SECONDARY OUTCOMES:
Rate of 2-year disease free survival | 2 years
  Disease free survival is calculated from the date of randomization to local recurrence, regional recurrence, distant metastasis or death. The rate of 2-year disease free survival is reported as the percentage of patients who are disease free survival for 2 years from the date of randomization.
Rate of 2-year overall survival | 2 years
  Overall survival is calculated from the date of randomization to death. The rate of 2-year overall survival is reported as the percentage of patients who are overall survival for 2 years from the date of randomization.
Health-related quality of life | 2 years
  Health-related quality of life will be measured and scored using the Chinese version of the University of Washington Quality of Life (UW-QOL) scale. Each score ranges from 0 to 100 points. The lower the score, the worse the functional perception.

CONTACTS AND LOCATIONS:
Overall Officials: Lai-ping Zhong, MD, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
After the completion of the trial.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years after completion of the trial, for 6 months.
Access Criteria: Data can be obtained upon scientifically sound request from the study PI, who will contact the Clinical Research Unit, Huashan Hospital, Fudan University. Access will be released after the approval from the Clinical Research Unit.